CLINICAL TRIAL: NCT07367789
Title: Prediction of Patient-reported Outcome Measure and Performance-based Measure After Total Knee Arthroplasty Using Instrumented Insoles and Deep Neural Networks
Brief Title: Prediction of Postoperative Outcomes After TKA Using Instrumented Insoles and DNN
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: GBIRB2025-324
Record Dates: First submitted 2025-12-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty
Keywords: Total knee arthroplasty; Prediction model; Deep neural network; Instrumented insole
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TKA Patients: Participants scheduled for primary unilateral total knee arthroplasty at either Yongin Severance Hospital or Gachon University Gil Medical Center. No intervention is assigned; all data are collected as part of observational evaluation.
  Interventions: Other: Instrumented Insole Gait Assessment

INTERVENTIONS:
Other: Instrumented Insole Gait Assessment — Participants undergo gait assessment using an instrumented insole system during the Timed Up and Go Test. The device is used solely for data collection and does not provide therapeutic intervention.

SUMMARY:
This multicenter prospective observational study aims to evaluate whether preoperative clinical variables and wearable sensor-derived gait features can predict postoperative improvement after total knee arthroplasty (TKA). Participants will undergo standardized gait assessments using instrumented insoles and complete validated patient-reported outcome measures (PROMs). Prediction models including linear regression, random forest, and deep neural networks will be applied and their performance compared.

DETAILED DESCRIPTION:
This study investigates predictive factors associated with postoperative improvement in both patient-reported outcomes and performance-based mobility measures among individuals undergoing total knee arthroplasty. Participants from two centers-Yongin Severance Hospital and Gachon University Gil Medical Center-will undergo preoperative collection of demographic data, body composition, muscle strength, comorbidity profiles, radiographic Kellgren-Lawrence grade, and wearable insole-derived gait data during the Timed Up and Go Test (TUGT). Postoperative outcomes at six weeks will include Western Ontario and McMaster Universities Arthritis Index (WOMAC) and TUGT.

Prediction models (linear regression, random forest, and deep neural network models) will be applied using consistent input variables. Model performance will be evaluated using accuracy and Receiver Operating Characteristic-Area Under the Curve (ROC-AUC). This study does not involve any therapeutic intervention and poses minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Diagnosed with knee osteoarthritis (Kellgren-Lawrence grade 1-4)
* Scheduled for primary Total Knee Arthroplasty (TKA) at either study site
* Able to walk independently on level ground (Functional Ambulation Categories, FAC ≥ 3)

Exclusion Criteria:

* Cancellation of scheduled TKA
* History of TKA on the same knee
* Neurological or musculoskeletal disorders affecting gait
* Pregnancy or possibility of pregnancy
* Any condition deemed inappropriate for study participation by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with knee osteoarthritis undergoing primary total knee arthroplasty at two hospitals in South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Improvement | Preoperative baseline; postoperative 6 weeks, 3 months, 6 months, and 12 months
  Improvement in patient-reported symptoms as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
  The WOMAC is a validated patient-reported outcome measure consisting of 24 items assessing pain (5 items), stiffness (2 items), and physical function (17 items). Each item is scored on a 5-point Likert scale (0-4), resulting in a total score ranging from 0 to 96, where higher scores indicate worse pain, stiffness, and functional limitation, and lower scores indicate better clinical status.
  Postoperative improvement is defined as a decrease of ≥15 points in the WOMAC total score compared with the preoperative baseline, corresponding to the minimal clinically important difference (MCID). Participants will be classified as "improved" or "not improved" based on this criterion (binary outcome).

SECONDARY OUTCOMES:
Timed Up and Go Test (TUGT) Improvement | Preoperative baseline; postoperative 6 weeks, 3 months, 6 months, and 12 months
  Improvement defined as a decrease in TUGT completion time from baseline (binary).

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srivastava AK; Surgical Management of Osteoarthritis of the Knee Work Group, Staff of the American Academy of Orthopaedic Surgeons. American Academy of Orthopaedic Surgeons Clinical Practice Guideline Summary of Surgical Management of Osteoarthritis of the Knee. J Am Acad Orthop Surg. 2023 Dec 15;31(24):1211-1220. doi: 10.5435/JAAOS-D-23-00338. Epub 2023 Oct 24. PMID 37883429
- [Background] Small SR, Bullock GS, Khalid S, Barker K, Trivella M, Price AJ. Current clinical utilisation of wearable motion sensors for the assessment of outcome following knee arthroplasty: a scoping review. BMJ Open. 2019 Dec 29;9(12):e033832. doi: 10.1136/bmjopen-2019-033832. PMID 31888943
- [Background] Ferreira AM, Salim R, Fogagnolo F, de Oliveira LFL, Riberto M, Kfuri M. The Value of a Standardized Knee Functional Assessment in Predicting the Outcomes of Total Knee Arthroplasty. J Knee Surg. 2022 Aug;35(10):1126-1131. doi: 10.1055/s-0040-1722321. Epub 2021 Jan 28. PMID 33511585
- [Background] Boekesteijn R, Smolders J, Busch V, Keijsers N, Geurts A, Smulders K. Objective monitoring of functional recovery after total knee and hip arthroplasty using sensor-derived gait measures. PeerJ. 2022 Sep 28;10:e14054. doi: 10.7717/peerj.14054. eCollection 2022. PMID 36193431
- [Background] Hsieh CY, Huang HY, Liu KC, Chen KH, Hsu SJ, Chan CT. Subtask Segmentation of Timed Up and Go Test for Mobility Assessment of Perioperative Total Knee Arthroplasty. Sensors (Basel). 2020 Nov 5;20(21):6302. doi: 10.3390/s20216302. PMID 33167444
- [Background] Salaffi F, Leardini G, Canesi B, Mannoni A, Fioravanti A, Caporali R, Lapadula G, Punzi L; GOnorthrosis and Quality Of Life Assessment (GOQOLA). Reliability and validity of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index in Italian patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2003 Aug;11(8):551-60. doi: 10.1016/s1063-4584(03)00089-x. PMID 12880577
- [Background] Tolk JJ, Janssen RPA, Prinsen CAC, Latijnhouwers DAJM, van der Steen MC, Bierma-Zeinstra SMA, Reijman M. The OARSI core set of performance-based measures for knee osteoarthritis is reliable but not valid and responsive. Knee Surg Sports Traumatol Arthrosc. 2019 Sep;27(9):2898-2909. doi: 10.1007/s00167-017-4789-y. Epub 2017 Nov 11. PMID 29128879
- [Background] Wilfong JM, Badley EM, Power JD, Gandhi R, Rampersaud YR, Perruccio AV. Discordance between self-reported and performance-based function among knee osteoarthritis surgical patients: Variations by sex and obesity. PLoS One. 2020 Jul 30;15(7):e0236865. doi: 10.1371/journal.pone.0236865. eCollection 2020. PMID 32730319
- [Background] Cooper NA, Rakel BA, Zimmerman B, Tonelli SM, Herr KA, Clark CR, Noiseux NO, Callaghan JJ, Sluka KA. Predictors of multidimensional functional outcomes after total knee arthroplasty. J Orthop Res. 2017 Dec;35(12):2790-2798. doi: 10.1002/jor.23596. Epub 2017 May 23. PMID 28471509
- [Background] Young-Shand KL, Dunbar MJ, Astephen Wilson JL. Individual Gait Features Are Associated with Clinical Improvement After Total Knee Arthroplasty. JB JS Open Access. 2020 Apr 6;5(2):e0038. doi: 10.2106/JBJS.OA.19.00038. eCollection 2020 Apr-Jun. PMID 33123659
- [Background] Batailler C, Lording T, De Massari D, Witvoet-Braam S, Bini S, Lustig S. Predictive Models for Clinical Outcomes in Total Knee Arthroplasty: A Systematic Analysis. Arthroplast Today. 2021 Apr 24;9:1-15. doi: 10.1016/j.artd.2021.03.013. eCollection 2021 Jun. PMID 33997202
- [Background] Olsen U, Lindberg MF, Rose C, Denison E, Gay C, Aamodt A, Brox JI, Skare O, Furnes O, Lee K, Lerdal A. Factors Correlated With Physical Function 1 Year After Total Knee Arthroplasty in Patients With Knee Osteoarthritis: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Jul 1;5(7):e2219636. doi: 10.1001/jamanetworkopen.2022.19636. PMID 35816307
- [Background] Harmelink KEM, Zeegers AVCM, Hullegie W, Hoogeboom TJ, Nijhuis-van der Sanden MWG, Staal JB. Are There Prognostic Factors for One-Year Outcome After Total Knee Arthroplasty? A Systematic Review. J Arthroplasty. 2017 Dec;32(12):3840-3853.e1. doi: 10.1016/j.arth.2017.07.011. Epub 2017 Aug 1. PMID 28927646
- [Background] Kluge F, Hannink J, Pasluosta C, Klucken J, Gassner H, Gelse K, Eskofier BM, Krinner S. Pre-operative sensor-based gait parameters predict functional outcome after total knee arthroplasty. Gait Posture. 2018 Oct;66:194-200. doi: 10.1016/j.gaitpost.2018.08.026. Epub 2018 Aug 24. PMID 30199778
- [Background] Berman AT, Quinn RH, Zarro VJ. Quantitative gait analysis in unilateral and bilateral total hip replacements. Arch Phys Med Rehabil. 1991 Mar;72(3):190-4. PMID 1998452
- [Background] Kramers-de Quervain IA, Stussi E, Muller R, Drobny T, Munzinger U, Gschwend N. Quantitative gait analysis after bilateral total knee arthroplasty with two different systems within each subject. J Arthroplasty. 1997 Feb;12(2):168-79. doi: 10.1016/s0883-5403(97)90063-2. PMID 9139099
- [Background] Feng Y, Liu Y, Fang Y, Chang J, Deng F, Liu J, Xiong Y. Advances in the application of wearable sensors for gait analysis after total knee arthroplasty: a systematic review. Arthroplasty. 2023 Oct 2;5(1):49. doi: 10.1186/s42836-023-00204-4. PMID 37779198
- [Background] Emmerzaal J, Corten K, van der Straaten R, De Baets L, Van Rossom S, Timmermans A, Jonkers I, Vanwanseele B. Movement Quality Parameters during Gait Assessed by a Single Accelerometer in Subjects with Osteoarthritis and Following Total Joint Arthroplasty. Sensors (Basel). 2022 Apr 12;22(8):2955. doi: 10.3390/s22082955. PMID 35458937
- [Background] Chatzaki C, Skaramagkas V, Kefalopoulou Z, Tachos N, Kostikis N, Kanellos F, Triantafyllou E, Chroni E, Fotiadis DI, Tsiknakis M. Can Gait Features Help in Differentiating Parkinson's Disease Medication States and Severity Levels? A Machine Learning Approach. Sensors (Basel). 2022 Dec 16;22(24):9937. doi: 10.3390/s22249937. PMID 36560313
- [Background] Moe-Nilssen R, Helbostad JL. Estimation of gait cycle characteristics by trunk accelerometry. J Biomech. 2004 Jan;37(1):121-6. doi: 10.1016/s0021-9290(03)00233-1. PMID 14672575
- [Background] Lee DW, Han HS, Lee MC, Ro DH. Prediction of postoperative gait speed change after bilateral primary total knee arthroplasty in female patients using a machine learning algorithm. Orthop Traumatol Surg Res. 2024 Nov;110(7):103842. doi: 10.1016/j.otsr.2024.103842. Epub 2024 Feb 19. PMID 38382881

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT07367789/Prot_SAP_000.pdf